CLINICAL TRIAL: NCT04305028
Title: Influence of Rivaroxaban 2.5 mg Two Times a Day for Intermittent Claudication and Exercise Tolerance in Patients With Symptomatic Peripheral Arterial Disease (PAD) - a Randomised Controlled Trial
Brief Title: Influence of Rivaroxaban for Intermittent Claudication and Exercise Tolerance in Patients With Symptomatic PAD
Acronym: PAD_RIV_CLI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Poznan University of Medical Sciences (Other)
Collaborators: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Other Study IDs: 132/20
Record Dates: First submitted 2020-03-09; First posted 2020-03-12 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease; Intermittent Claudication; Rivaroxaban
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication | interventions — Rivaroxaban; Aspirin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood -EDTA samples, Serum samples, DNA samples
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental: Rivaroxaban [2.5 mg] + Aspirin: Drug: Rivaroxaban 2.5 mg twice daily, tablet Drug: Aspirin 75-100 mg once daily, tablet
  Interventions: Drug: Rivaroxaban; Drug: Aspirin
- Active Comparator: Aspirin: Drug: Aspirin 75-100 mg once daily, tablet
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Rivaroxaban — Rivaroxaban 2.5 MG (Xarelto) twice daily, tablet
  Other Names: Rivaroxaban 2.5 MG; Xarelto
  Groups: Experimental: Rivaroxaban [2.5 mg] + Aspirin
Drug: Aspirin — Aspirin 75-100 mg once daily, tablet
  Other Names: Acetylsalicylic acid

SUMMARY:
The aim of the conducted research is to evaluate the protective effect of rivaroxaban (trade name of the Xarelto medicinal product), administered together with acetylsalicylic acid (ASA), in comparison with the effectiveness of using ASA alone, in relation to the distance of claudication and exercise tolerance in patients with PAD over a period of 3 months. At present, COMPASS results show that rivaroxaban vascular dose (2.5 mg twice daily) in combination with ASA (75-100 mg once daily) provides more effective cardiovascular protection (defined as cardiovascular death, vascular, myocardial infarction and stroke) compared to ASA alone. So far, however, no scientific studies have been carried out into account the effect of the drug on the progress of PAD and exercise tolerance in patients.

DETAILED DESCRIPTION:
EXISTING KNOWLEDGE AND MAIN ASSUMPTIONS OF THE PROJECT.

Atherosclerosis is the most common cause of peripheral artery disease (PAD). The first symptom of PAD is intermittent claudication (IC), which is characterized by the occurrence of pain, cramps, numbness, and discomfort in the lower limb muscles. They gradually intensify while walking, forcing the patient to stop. The symptoms are caused by continuous, specific physical effort and quickly disappear when it is stopped. The reduction of the possibility of walking leads to a decrease in the quality of life of patients and adds to other dangerous consequences of atherosclerosis, increased risk of cardiovascular incidents (myocardial infarction (MI), stroke, acute lower limb ischemia, Micker M et al. 2006).

Pharmacological treatment of patients with IC is aimed at modifying cardiovascular risk factors and improving the quality of life by alleviating pain and prolonging the claudication distance (Goszcz et al., 2009).

1. New possibilities for the pharmacotherapy of patients with symptomatic PAD.

   According to the adopted TASC (The Trans Atlantic Inter-Society Consensus), and its TASC II supplement concerning aspects of management and treatment of patients with chronic limb ischemia (CLI), drugs used in PAD are divided into nine groups: those with documented clinical effect used in IC (cilostazol and naphthydrofuryl), drugs with probable clinical effect used in IC (carnitine and propyl-L-carnitine), lipid-lowering drugs (statins), drugs with insufficiently proven clinical effects (penthoxyphilin), anticoagulants, L-arginine, 5-hydroxytryptamine (ketanserin) antagonism, buflomedil, and defibrotide.
2. Antiplatelet drugs

   Antiplatelet drugs are used to prevent thrombotic complications in the course of myocardial infarction, stroke, and thrombi in peripheral arteries. Acetylsalicylic acid (ASA, aspirin) at doses of 75-325 mg per day, ticlopidine at doses of 250 mg twice a day, and clopidogrel at doses of 75 mg once a day (CAPRIE, 1996) are proven to be effective in PAD patients. Recently there have been reports of beneficial effects of policosanol (a cholesterol-lowering drug with an antiplatelet effect), which prolongs the claudication distance after 10 weeks of treatment (10 mg once a day; clinical trial). The results of ASA (100 mg daily) were however inconclusive (Illnait et al., 2008).

   The group of new antiplatelet drugs, used in PAD patients, includes rivaroxaban (trade name Xarelto), which in a vascular dose (2.5 mg twice a day) combined with ASA (75-100 mg once a day) provides more effective cardiovascular protection (defined together as cardiovascular death, MI and stroke) compared to ASA alone in the COMPASS study (Anand SS et al. 2018; Olinic DM et al. 2018; Connolly SJ, 2018).

   Other studies with the acronyms MACE and MALE, conducted in the PAD patients of nearly 5,000 cases in total, confirm that the use of rivaroxaban provides comprehensive vascular protection in PAD. The former showed a 28% reduction in the risk of cardiovascular death/myocardial infarction/brain stroke, the latter a 44% reduction in the risk of acute lower limb ischemia and a 46% reduction in the risk of acute/chronic limb ischemia and a 70% reduction in the risk of large amputations. This is the only anticoagulant that, in combination with ASA, reduces mortality in patients with coronary artery disease (CAD) and PAD. At the same time, Xarelto, in a vascular dose, in combination with ASA, does not cause a significant increase in the risk of major bleedings compared to ASA itself. So far, this drug has not been tested in the context of prolongation of the claudication distance.

   Rivaroxaban inhibits the formation of thrombin and clots by directly inhibiting factor Xa (activated factor X), thus preventing the transformation of prothrombin into thrombin and interrupting the final common path of the blood clotting cascade. This drug competitively inhibits factor Xa with 10,000 times the selectivity of related serine proteases such as thrombin and factors VIIa, IXa, and XIa. Numerous experimental data suggest the role of clotting system components in regulating atherosclerosis progression (Borensztajn K et al., 2008; Borissoff et al., 2009; Platek and Szymanski, 2019). Various factors of the coagulation cascade mediate these activities, and the broadest spectrum of action concerns the effect of the complex of factor Xa and thrombin precisely.

   Scientific research confirms the pleiotropic effects of rivaroxaban on the cardiovascular system. However, most of the currently available observations come from basic research whose results need to be confirmed in clinical trials. Among the planned clinical trials that may establish pleiotropic rivaroxaban actions, the PRE -FER-AF study (PREvention oF thromboembolic events - European Registry in Atrial Fibrillation) is mentioned as the most important. This study aims to determine the efficacy of oral anticoagulants other than vitamin K antagonists (NOAC) in preventing endothelial dysfunction and atherosclerosis progression in patients with atrial fibrillation. However, it will not provide information on the effect of the drug on the progress of PAD or exercise tolerance.
3. The objective

   The aim of the study is to assess the protective efficacy of rivaroxaban, administered together with ASA, in comparison with the efficacy of ASA alone, with respect to intermittent claudication and exercise tolerance in patients with PAD over a 3-month period.
4. Type of study

   Prospective, observational, unblinded (open), randomized, case-control, single-centre.
5. Description of the study group (age, gender, health status, size of the group).

   The study will include PAD patients in Fountaine stage II, hospitalized in the Clinical Hospital of Transfiguration (Department of Vascular and Endovascular Surgery, Angiology and Phlebology of the Poznan University of Medical Sciences), monitored in the adjacent Outpatient Clinic or referred by cooperating physicians who will use a different protocol of anticoagulation pharmacotherapy to prevent thrombotic events. The recommended pharmacotherapy does not exceed the standard of treatment in patients with PAD.

   5.1 Size of the study group. At least 60 PAD patients will be included. The collection and observation of the study group will take place until the scientific goal of the study is achieved. Therefore the possibility of increasing the recruitment of patients for the study is assumed up to 100 patients.

   5.2 Characteristics of the study group. The inclusion/exclusion criteria, medical history, and cardiovascular risk factors will be examined. Then patients will be subjected to objective assessment of exercise tolerance, assessment of claudication distance, implementation of anticoagulation pharmacotherapy protocol and prospective study protocol. Venous blood samples (9-18 ml), and capillary blood for diagnostic, biochemical, and molecular analysis will be collected. Costs will be shared between cooperating centers.

   5.3 Pharmacotherapy. Vascular doses of drugs will be used in one group: 1 x/day ASA 75-100 mg and in the other: 1 x/day ASA 75-100 mg + 2 x/day 2.5 mg Xarelto.
6. Methods The general study plan assumes up to 5 visits of the patient to the cooperating centers during the study. First visit to the Hospital-Outpatient Clinic for recruitment (interview with the patient, obtaining written consent, patient registration, the appointment of the next visit, and optionally USG-Doppler of arteries). Second visit to the hospital's blood collection point for fasting blood tests (blood collection for tests and optionally USG-Doppler of arteries). During the third and fourth visits at University of Physical Education treadmill tests with additional tests (ECG, ABI, TCPO2 measurements before and after treadmill test, as well as biochemical evaluation of effort tolerance and subjective assessment of effort using Borg scale) will be performed. During third visit, randomization will also be done. The fourth visit will be scheduled after three months. Then data will be collected and analyzed. During the fifth visit, USG-Doppler of arteries will be performed, and a patient recommendation will be issued.

6.1 Clinical characteristics of the studied population. The following clinical data will be collected for the study: a) results of aortic and lower limb arteries imaging, b) results of heart function tests, c) assessment of the occurrence and severity of atherosclerotic lesions in blood vessels (including: ABI, IMT,TcPO2 value), d) results of fasting venous blood laboratory tests including blood lipid parameters, glucose metabolism, liver and renal function, homocysteine, folic acid, peripheral blood morphology, blood coagulation parameters, e) blood pressure parameters, f) results of virological and bacteriological tests, g) anthropometric data, h) smoking status, i) pharmacotherapy j) coexisting diseases, k) pain, l) family history of cardiovascular disease and cancer.

6.2 Treadmill test. The effect of pharmacotherapy will be assessed based on the treadmill test that will be carried out according to Gardner protocol (Gardner et al., 1991). Patients will march on a treadmill at a constant speed of 3.2 km/h. The initial angle of the slope will be 0% and will be raised by 2% every 2 minutes. The test will be carried out in the Laboratory of Functional Testing of the Department of Physiology and Biochemistry of the University of Physical Education in Poznan, with no contraindications (based on the result of an ECG). The subjects will be tested at each of the test dates to assess the claudication distance on the Katana S30p medical treadmill (Lode BV, Netherlands) (Mika et al. 2009). The total time of each test will not exceed 16 minutes 40 seconds, and the regeneration time will be at least 5 minutes. When the patient reports pain (i.e., grade 2 on a subjective pain assessment scale), the time of occurrence of the claudication will be recorded, from which the claudication distance (DGCH) will be estimated. The test will be interrupted when very severe pain occurs that prevents further walking (step 5 corresponding to maximum walking time), and the maximum walking time will then be recorded. The maximum walking time will be used to estimate the maximum walking distance (DGMAX). Once the treadmill tests have been completed, patients will undergo a control ECG examination to exclude ischemic changes in the heart muscle and cardiac arrhythmias.

6.3. Evaluation of exercise tolerance. The assessment of exercise tolerance will be carried out based on the duration of the effort and questionnaires (Borg scale; Smarż et al. 2015), and biochemical exponents (metabolic equivalent MET-s will be estimated; Bires AM et al., 2013). At rest and 3 minutes after the exercise, the intensity of metabolic exercise acidosis will be assessed based on lactate concentration in capillary blood taken from the fingertip. At the same time, venous blood will also be collected for other biochemical tests, including gasometry.

6.4 Length of observation. The effects of the treatment will be assessed within three months, but the observation period can be extended to a maximum of 12 months.

6.5 End points of the study. The main endpoints of this study and the complications have been developed in accordance with the results adopted in the COMPASS study. Parameters related to the effects of the treadmill test were added.

6.6 Biological material and its use. Blood samples will be collected for further analysis and DNA extraction. The concentration of lactate will be tested using EDGE Blood Lactate Test Strip, ApexBio, (Taiwan). The level of selected blood biomarkers will be assessed by the immunoenzymatic method (ELISA) for proteins, and TaqMan tests or corresponding methods for circulating miRNAs and DNA.

ELIGIBILITY:
Inclusion Criteria:

1. PAD, the Fontaine classification II

Exclusion Criteria:

1. Severe heart failure with known ejection fraction <30% or NYHA class III or IV symptoms
2. High risk of bleeding
3. Stroke with one month or any history of hemorrhaging or lacunar stroke
4. Estimated glomerular filtration rate <15 ml/ml
5. Need for dual antiplatelet therapy, other non-aspirin antiplatelet therapy/, oral anticoagulant therapy/
6. The known non-cardiovascular disease that is associated with poor prognosis (i.n, metastatic cancer)
7. History of hypersensitivity or known contraindication for rivaroxaban, aspirin
8. Systemic treatment with strong inhibitors of CYP 3A4 as well as p-glycoprotein or strong inducers of CYP 3M
9. Any known hepatic disease associated with coagulopathy
10. Concurrent participation in another study with an investigational drug
11. Known contraindication to any study-related procedures* Concerns: Absolute contraindications to an exercise test
12. Respiratory failure
13. BMI above or equal 40
14. Musculoskeletal dysfunction preventing walking (e.g. amputations)

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The primary selection criterion for all respondents is the presence of PAD and the Caucasian ancestry. PAD patients with intermittent claudication and no clinical contraindications to the treadmill test will be enrolled in the study. Patients with PAD in Stage II Fountaine will be qualified for the study. The disease will be confirmed with an ankle-brachial index (ABI), with a result of less than 0.90. For all participants, ABI will be measured at the beginning of the study; the result will be calculated from the ratio of the highest systolic blood pressure on the limb to the highest systolic blood pressure on the shoulder.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-03-10 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Diagnosed with Stroke at 3 Months | 3 months
  Number of participants diagnosed with ischemic or hemorrhagic stroke
Number of Participants Diagnosed with Myocardial Infarction (MI) at 3 Months | 3 months
  Number of participants diagnosed with myocardial infarction
Number of Participants who Died from Cardiovascular Causes at 3 Months | 3 months
  Number of participants who died because of Cardiovascular causes
Number of Participants who Died from Any Cause at 3 Months | 3 months
  Number of Participants who died for any reason not related to accidents.
Number of Participants Diagnosed with Acute Limb Ischaemia (ALI) at 3 Months | 3 months
  Number of participants diagnosed with acute limb ischaemia definied as limb threatening ischaemia with evidence of acute arterial obstruction by radiological criteria or a new pulse deficit leading to an intervention (ie, surgery, thrombolysis, peripheral angioplasty, or amputation.
Number of Participants Diagnosed with Major Limb Amputation (AMI) at 3 Months | 3 months
  Number of participants diagnosed with major limb amputation defined as amputations due to a vascular event above the forefoot, or defined as minor amputation if involving the forefoot and digits.
Change From Baseline in the Distance of Intermittent Claudication (Δ Dch) at 3 Months | 3 months
  Change in the distance of intermittent claudication in the test according to Gardner's protocol
Change From Baseline in the Maximal Distance of Intermittent Claudication (Δ Dmax) at 3 Months | 3 months
  Change in the maximal distance of intermittent claudication in the test according to Gardner's protocol

OTHER OUTCOMES:
Number of Participants Diagnosed with Fatal Bleeding (FB) at 3 Months | 3 months
  Number of participants diagnosed with bleeding that directly results in death within 7 days after its occurrence
Number of Participants Diagnosed with Non-Fatal Symptomatic Intracranial Haemorrhage (IH) at 3 Months | 3 months
  Number of participants diagnosed with non-fatal symptomatic intracranial haemorrhage.
Number of Participants Diagnosed with Non-Fatal, Non-Intracranial Haemorrhage (Non-IH) Symptomatic Bleeding at 3 Months into a critical organ | 3 months
  Number of participants diagnosed with non-fatal, non-intracranial haemorrhage symptomatic bleeding into a critical organ
Number of Participants Diagnosed with Other Major Bleeding at 3 Months | 3 months
  Number of participants diagnosed with other major bleeding defined as surgical site bleeding, surgical site bleeding, that requires reoperation or bleeding leading to hospitalization
Number of Participants Diagnosed with Fatal or Symptomatic Bleeding into a Critical Organ at 3 Months | 3 months
  Number of participants diagnosed with fatal or symptomatic bleeding into a critical organ
Number of Participants Diagnosed with Major Bleeding according to ISTH criteria at 3 Months | 3 months
  Number of participants diagnosed with major bleeding according to modified the International Society on Thrombosis and Haemostasis (ISTH) criteria for major bleeding, defined as the composite of bleeding that was fatal, symptomatic bleeding into a critical organ, surgical site requiring reoperation, or requiring hospitalization (including presentation to an acute care facility without an overnight stay).(ISTH)/Scientific and Standardization Committee (SSC) definitions
Number of Participants Diagnosed with Minor Bleeding at 3 Months | 3 months
  Number of participants diagnosed with clinically relevant minor bleeding defined as an acute or subacute clinically overt bleed that does not meet the criteria for a major bleed but prompts a clinical response, in that it leads to at least one of the following: 1) a hospital admission for bleeding, or 2) a physician-guided medical or surgical treatment for bleeding, or 3) a change in antithrombotic therapy (including interruption or discontinuation of study drug).
Number of Participants Diagnosed with Gastrointestinal Bleeding at 3 Months | 3 months
  Number of participants diagnosed with gastrointestinal bleeding.
Number of Participants Diagnosed with Intracranial Bleeding at 3 Months | 3 months
  Number of participants diagnosed with intracranial bleeding
Number of Participants Diagnosed with Genitourinary Bleeding at 3 Months. | 3 months
  Number of participants diagnosed with genitourinary bleeding.
Number of Participants Diagnosed with Ocular Bleeding at 3 Months. | 3 months
  Number of participants diagnosed with ocular bleeding.
Number of Participants Diagnosed with Skin Bleeding at 3 Months. | 3 months
  Number of participants diagnosed with skin bleeding.
Number of Participants Diagnosed with Respiratory Bleeding at 3 Months. | 3 months
  Number of participants diagnosed with respiratory bleeding.
Number of Participants Diagnosed with Other Bleeding at 3 Months. | 3 months
  Number of participants diagnosed with bleeding other than: gastrointestinal, intracranial, genitourinary, ocular, skin, respiratory.

CONTACTS AND LOCATIONS:
Overall Officials: Zbigniew Krasiński, Prof, MD, Principal Investigator — Poznan University of Medical Sciences; Ewa Strauss, PhD, Study Director — Poznan University of Medical Sciences

IPD SHARING:
Plan to Share IPD: Undecided
These data will be made available on reasonable request

REFERENCES:
- [Result] Anand SS, Bosch J, Eikelboom JW, Connolly SJ, Diaz R, Widimsky P, Aboyans V, Alings M, Kakkar AK, Keltai K, Maggioni AP, Lewis BS, Stork S, Zhu J, Lopez-Jaramillo P, O'Donnell M, Commerford PJ, Vinereanu D, Pogosova N, Ryden L, Fox KAA, Bhatt DL, Misselwitz F, Varigos JD, Vanassche T, Avezum AA, Chen E, Branch K, Leong DP, Bangdiwala SI, Hart RG, Yusuf S; COMPASS Investigators. Rivaroxaban with or without aspirin in patients with stable peripheral or carotid artery disease: an international, randomised, double-blind, placebo-controlled trial. Lancet. 2018 Jan 20;391(10117):219-229. doi: 10.1016/S0140-6736(17)32409-1. Epub 2017 Nov 10. PMID 29132880
- [Result] Borensztajn K, Peppelenbosch MP, Spek CA. Factor Xa: at the crossroads between coagulation and signaling in physiology and disease. Trends Mol Med. 2008 Oct;14(10):429-40. doi: 10.1016/j.molmed.2008.08.001. Epub 2008 Sep 4. PMID 18774340
- [Result] Borissoff JI, Spronk HM, Heeneman S, ten Cate H. Is thrombin a key player in the 'coagulation-atherogenesis' maze? Cardiovasc Res. 2009 Jun 1;82(3):392-403. doi: 10.1093/cvr/cvp066. Epub 2009 Feb 19. PMID 19228706
- [Result] Bires AM, Lawson D, Wasser TE, Raber-Baer D. Comparison of Bruce treadmill exercise test protocols: is ramped Bruce equal or superior to standard bruce in producing clinically valid studies for patients presenting for evaluation of cardiac ischemia or arrhythmia with body mass index equal to or greater than 30? J Nucl Med Technol. 2013 Dec;41(4):274-8. doi: 10.2967/jnmt.113.124727. Epub 2013 Nov 12. PMID 24221922
- [Result] CAPRIE Steering Committee. A randomised, blinded, trial of clopidogrel versus aspirin in patients at risk of ischaemic events (CAPRIE). CAPRIE Steering Committee. Lancet. 1996 Nov 16;348(9038):1329-39. doi: 10.1016/s0140-6736(96)09457-3. PMID 8918275
- [Result] Connolly SJ, Eikelboom JW, Bosch J, Dagenais G, Dyal L, Lanas F, Metsarinne K, O'Donnell M, Dans AL, Ha JW, Parkhomenko AN, Avezum AA, Lonn E, Lisheng L, Torp-Pedersen C, Widimsky P, Maggioni AP, Felix C, Keltai K, Hori M, Yusoff K, Guzik TJ, Bhatt DL, Branch KRH, Cook Bruns N, Berkowitz SD, Anand SS, Varigos JD, Fox KAA, Yusuf S; COMPASS investigators. Rivaroxaban with or without aspirin in patients with stable coronary artery disease: an international, randomised, double-blind, placebo-controlled trial. Lancet. 2018 Jan 20;391(10117):205-218. doi: 10.1016/S0140-6736(17)32458-3. Epub 2017 Nov 10. PMID 29132879
- [Result] Gardner AW, Skinner JS, Cantwell BW, Smith LK. Progressive vs single-stage treadmill tests for evaluation of claudication. Med Sci Sports Exerc. 1991 Apr;23(4):402-8. PMID 2056896
- [Result] Goszcz A, Woroń J, Kostka-Trąbka E. Farmakoterapia przewlekłego niedokrwienia kończyn dolnych (PAD). [Pharmacotherapy for chronic lower limb ischaemia (PAD)] Farm Współ 2009; 2: 91-96.
- [Result] Illnait J, Castano G, Alvarez E, Fernandez L, Mas R, Mendoza S, Gamez R. Effects of policosanol (10 mg/d) versus aspirin (100 mg/d) in patients with intermittent claudication: a 10-week, randomized, comparative study. Angiology. 2008 Jun-Jul;59(3):269-77. doi: 10.1177/0003319707306963. Epub 2008 Apr 2. PMID 18388038
- [Result] Micker M, Chęciński P, Synowiec T. Postępowanie w przewlekłym niedokrwieniu kończyn dolnych.[Treatment of chronic ischaemia in the lower extremitie] Przew Lek 2006; 5: 12-21.
- [Result] Mika P, Spannbauer A, Cencora A. Zmiana wzorca chodu i dystansu marszu w trakcie zapoznawania się pacjenta z chromaniem przestankowym ze specyfiką marszu na bieżni. [Change of the walking pattern and walking distance during the patient's acquaintance with the diaphragm cladication on the treadmill] Pielęg Chir Angiol 2009; 2: 65-69.
- [Result] Olinic DM, Tataru DA, Homorodean C, Spinu M, Olinic M. Antithrombotic treatment in peripheral artery disease. Vasa. 2018 Feb;47(2):99-108. doi: 10.1024/0301-1526/a000676. Epub 2017 Nov 21. PMID 29160765
- [Result] Płatek AE, Szymański FM. Riwaroksaban - nowy lek plejotropowy o szerokim spektrum działań [Riwaroxaban - a new broad spectrum pleiotropic drug] Choroby Serca i Naczyń 2019, tom 16, nr 1, 34-40,
- [Result] Pocock SJ, Simon R. Sequential treatment assignment with balancing for prognostic factors in the controlled clinical trial. Biometrics. 1975 Mar;31(1):103-15. PMID 1100130
- [Result] Smarż K, Jaxa-Chamiec T, Budaj A. Metody oceny wydolności fizycznej pacjentów kardiologicznych - elektrokardiograficzny, spiroergometryczny i echokardiograficzny test wysiłkowy. [Methods of assessing physical fitness of cardiac patients - electrocardiographic, spiroergometric and echocardiographic exercise test.] Postępy Nauk Medycznych, t. XXVIII, nr 11B, 2015
- [Result] Taves DR. Minimization: a new method of assigning patients to treatment and control groups. Clin Pharmacol Ther. 1974 May;15(5):443-53. doi: 10.1002/cpt1974155443. No abstract available. PMID 4597226
- See also: Xarelto description — http://leki.urpl.gov.pl/files/Xarelto.pdf

DOCUMENTS (3):
  • Study Protocol (2020-02-13): https://cdn.clinicaltrials.gov/large-docs/28/NCT04305028/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-13): https://cdn.clinicaltrials.gov/large-docs/28/NCT04305028/SAP_001.pdf
  • Informed Consent Form (2020-02-13): https://cdn.clinicaltrials.gov/large-docs/28/NCT04305028/ICF_002.pdf